CLINICAL TRIAL: NCT04756115
Title: Impact of Nutritional and Inflammatory Status in Patients With Critical Limb-threatening Ischemia: a Retrospective Cohort Stud
Brief Title: Impact of Nutritional and Inflammatory Status in Patients With Critical Limb-threatening Ischemia
Status: Completed | Type: Observational
Sponsor: Vascular Investigation Network Spanish Society for Angiology and Vascular Surgery (Network)
Collaborators: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Sponsor
Other Study IDs: PNI-2016/19
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Critical Lower Limb Ischemia; Postoperative Complications
Keywords: Peripheral Arterial Disease; Critical Limb Ischemia; Biomarkers; Prognostic Nutritional Index; Mortality Rate
MeSH Terms: conditions — Postoperative Complications; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia | interventions — Vascular Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CASES: Adults (age<18 years) diagnosed with a first episode of critical limb ischemia revascularized at our center from January 2016 to July 2019.
  Interventions: Procedure: Vascular Surgery.

INTERVENTIONS:
Procedure: Vascular Surgery. — Open Vascular, endovascular or hybrid procedures.

SUMMARY:
The peripheral arterial disease (PAD) has been associated with all-cause and cardiovascular mortality. Despite minimally invasive endovascular techniques, patients with critical limb-threatening ischemia (CLTI) have a poor prognosis with a high mortality that is comparable that of cancer.

The inflammatory activity has a crucial role for the development and prognosis of atherosclerosis. Recently, different inflammatory biomarkers such as the neutrophil to lymphocyte ratio (NLR), platelet to lymphocyte ratio (PLR) and lymphocyte to monocyte ratio (LMR) have been associated with severity and prognosis in patients with PAD.

Additionally, patients with CLTI present several independent risk factors for malnutrition. For this reason, malnutrition represents an independent risk factor for mortality and post-operative complications. In this context, the Prognostic Nutritional Index (PNI) associates the nutritional and inflammatory status of patients.

This study shows the clinical applicability of the different pre-operative nutritional and inflammatory biomarkers in patients with CLTI. This study does not collect any patient identifiable information.

DETAILED DESCRIPTION:
In order to show the relevance of patient's inflammatory status regarding the prognosis of PAD, this study establishes the correlation between pre-operative pro-inflammatory biomarkers represented by NLR, LMR and PLR with short-term mortality and major amputations at 6-months. Likewise, the association between the pre-operative PNI with short-term mortality and major amputation at 6-months revealing the impact of nutritional status.

- Data Collection: Demographic and clinical data. The initial surgical technique. The peri-operative outcomes Mortality and major amputation. The hemogram and biochemistry analysis were recorded preoperatively, at 48-hours after admission The inflammatory state was measured by the ratios of neutrophil/lymphocyte (NLR), lymphocyte/monocyte (LMR) and platelet/lymphocyte (PLR).

The nutritional status was estimated by the PNI = (serum albumin g/dL x 10) + (lymphocytes/μL + 0.005).

- Statistical Analysis: significant values p<0.05. Descriptive analysis was presented as mean values and respective standard deviations.

The chi-squared test and Student t-test were used for variables that followed a normal distribution.

A non-parametric test was performed for the rest of variables (Mann-Whitney U). Spearman and Pearson correlations coefficients were calculated to determine the association between biomarkers and the hospital length-of-stay.

For the multivariate analysis a logistic regression was performed. A receiver operating characteristic (ROC) curve analysis was applied to establish a cut-off point with the corresponding area under the curve (AUC), 95% confidence interval (95%CI), sensitivity (S) and specificity (E) for short-term mortality and major amputation at six months.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with a first episode of critical limb ischemia revascularized at our center from January 2016 to July 2019.

Exclusion Criteria:

* Patients with acute limb ischaemia.
* Patients with CLTI revascularized before 2016.
* Patients without serum albumin collected in the first 48 hours after admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a first episode of critical limb ischemia revascularized.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
6-month mortality | 6-month
  Correlation between pre-operative pro-inflammatory and nutritional biomarkers with mortality after vascular surgery.

SECONDARY OUTCOMES:
6-month major amputation | 6-month
  Correlation between pre-operative pro-inflammatory and nutritional biomarkers with major amputation after vascular surgery.

OTHER OUTCOMES:
Hospital length-of-stay | Immediately after the surgery
  Correlation between pre-operative pro-inflammatory and nutritional biomarkers with hospital length-of-stay after vascular surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Resnick HE, Lindsay RS, McDermott MM, Devereux RB, Jones KL, Fabsitz RR, Howard BV. Relationship of high and low ankle brachial index to all-cause and cardiovascular disease mortality: the Strong Heart Study. Circulation. 2004 Feb 17;109(6):733-9. doi: 10.1161/01.CIR.0000112642.63927.54. PMID 14970108
- [Result] Ankle Brachial Index Collaboration; Fowkes FG, Murray GD, Butcher I, Heald CL, Lee RJ, Chambless LE, Folsom AR, Hirsch AT, Dramaix M, deBacker G, Wautrecht JC, Kornitzer M, Newman AB, Cushman M, Sutton-Tyrrell K, Fowkes FG, Lee AJ, Price JF, d'Agostino RB, Murabito JM, Norman PE, Jamrozik K, Curb JD, Masaki KH, Rodriguez BL, Dekker JM, Bouter LM, Heine RJ, Nijpels G, Stehouwer CD, Ferrucci L, McDermott MM, Stoffers HE, Hooi JD, Knottnerus JA, Ogren M, Hedblad B, Witteman JC, Breteler MM, Hunink MG, Hofman A, Criqui MH, Langer RD, Fronek A, Hiatt WR, Hamman R, Resnick HE, Guralnik J, McDermott MM. Ankle brachial index combined with Framingham Risk Score to predict cardiovascular events and mortality: a meta-analysis. JAMA. 2008 Jul 9;300(2):197-208. doi: 10.1001/jama.300.2.197. PMID 18612117
- [Result] Varu VN, Hogg ME, Kibbe MR. Critical limb ischemia. J Vasc Surg. 2010 Jan;51(1):230-41. doi: 10.1016/j.jvs.2009.08.073. PMID 20117502
- [Result] Hirsch AT, Hartman L, Town RJ, Virnig BA. National health care costs of peripheral arterial disease in the Medicare population. Vasc Med. 2008 Aug;13(3):209-15. doi: 10.1177/1358863X08089277. PMID 18687757
- [Result] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). J Vasc Surg. 2007 Jan;45 Suppl S:S5-67. doi: 10.1016/j.jvs.2006.12.037. No abstract available. PMID 17223489
- [Result] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH; GVG Writing Group. Global vascular guidelines on the management of chronic limb-threatening ischemia. J Vasc Surg. 2019 Jun;69(6S):3S-125S.e40. doi: 10.1016/j.jvs.2019.02.016. Epub 2019 May 28. PMID 31159978
- [Result] Stamler J, Stamler R, Neaton JD, Wentworth D, Daviglus ML, Garside D, Dyer AR, Liu K, Greenland P. Low risk-factor profile and long-term cardiovascular and noncardiovascular mortality and life expectancy: findings for 5 large cohorts of young adult and middle-aged men and women. JAMA. 1999 Dec 1;282(21):2012-8. doi: 10.1001/jama.282.21.2012. PMID 10591383
- [Result] Vidula H, Tian L, Liu K, Criqui MH, Ferrucci L, Pearce WH, Greenland P, Green D, Tan J, Garside DB, Guralnik J, Ridker PM, Rifai N, McDermott MM. Biomarkers of inflammation and thrombosis as predictors of near-term mortality in patients with peripheral arterial disease: a cohort study. Ann Intern Med. 2008 Jan 15;148(2):85-93. doi: 10.7326/0003-4819-148-2-200801150-00003. PMID 18195333
- [Result] Paquissi FC. The role of inflammation in cardiovascular diseases: the predictive value of neutrophil-lymphocyte ratio as a marker in peripheral arterial disease. Ther Clin Risk Manag. 2016 May 27;12:851-60. doi: 10.2147/TCRM.S107635. eCollection 2016. PMID 27313459
- [Result] Demirdal T, Sen P. The significance of neutrophil-lymphocyte ratio, platelet-lymphocyte ratio and lymphocyte-monocyte ratio in predicting peripheral arterial disease, peripheral neuropathy, osteomyelitis and amputation in diabetic foot infection. Diabetes Res Clin Pract. 2018 Oct;144:118-125. doi: 10.1016/j.diabres.2018.08.009. Epub 2018 Sep 1. PMID 30176260
- [Result] Correia MI, Waitzberg DL. The impact of malnutrition on morbidity, mortality, length of hospital stay and costs evaluated through a multivariate model analysis. Clin Nutr. 2003 Jun;22(3):235-9. doi: 10.1016/s0261-5614(02)00215-7. PMID 12765661
- [Result] Buzby GP, Mullen JL, Matthews DC, Hobbs CL, Rosato EF. Prognostic nutritional index in gastrointestinal surgery. Am J Surg. 1980 Jan;139(1):160-7. doi: 10.1016/0002-9610(80)90246-9. PMID 7350839
- [Result] Chen QJ, Qu HJ, Li DZ, Li XM, Zhu JJ, Xiang Y, Li L, Ma YT, Yang YN. Prognostic nutritional index predicts clinical outcome in patients with acute ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention. Sci Rep. 2017 Jun 12;7(1):3285. doi: 10.1038/s41598-017-03364-x. PMID 28607442
- [Result] Teker Acikel ME, Korkut AK. Impact of Controlling Nutritional Status Score (CONUT) and Prognostic Nutritional Index (PIN) on Patients Undergoing Coronary Artery Bypass Graft Surgery. Heart Surg Forum. 2019 Jul 25;22(4):E294-E297. doi: 10.1532/hsf.2493. PMID 31398095
- [Result] Salomon du Mont L, Leclerc B, Morgant MC, Besch G, Laubriet A, Steinmetz E, Rinckenbach S. Impact of Nutritional State on Critical Limb Ischemia Early Outcomes (DENUCRITICC Study). Ann Vasc Surg. 2017 Nov;45:10-15. doi: 10.1016/j.avsg.2017.04.030. Epub 2017 May 8. PMID 28495537
- [Result] van Stijn MF, Korkic-Halilovic I, Bakker MS, van der Ploeg T, van Leeuwen PA, Houdijk AP. Preoperative nutrition status and postoperative outcome in elderly general surgery patients: a systematic review. JPEN J Parenter Enteral Nutr. 2013 Jan;37(1):37-43. doi: 10.1177/0148607112445900. Epub 2012 May 1. PMID 22549764
- [Result] Bozzetti F, Gianotti L, Braga M, Di Carlo V, Mariani L. Postoperative complications in gastrointestinal cancer patients: the joint role of the nutritional status and the nutritional support. Clin Nutr. 2007 Dec;26(6):698-709. doi: 10.1016/j.clnu.2007.06.009. Epub 2007 Aug 1. PMID 17683831
- [Result] Owens CD, Kim JM, Hevelone ND, Gasper WJ, Belkin M, Creager MA, Conte MS. An integrated biochemical prediction model of all-cause mortality in patients undergoing lower extremity bypass surgery for advanced peripheral artery disease. J Vasc Surg. 2012 Sep;56(3):686-95. doi: 10.1016/j.jvs.2012.02.034. Epub 2012 May 2. PMID 22554422
- [Result] Peacock MR, Farber A, Eslami MH, Kalish JA, Rybin D, Doros G, Shah NK, Siracuse JJ. Hypoalbuminemia Predicts Perioperative Morbidity and Mortality after Infrainguinal Lower Extremity Bypass for Critical Limb Ischemia. Ann Vasc Surg. 2017 May;41:169-175.e4. doi: 10.1016/j.avsg.2016.08.043. Epub 2017 Feb 27. PMID 28242402
- [Result] Stabile E, Kinnaird T, la Sala A, Hanson SK, Watkins C, Campia U, Shou M, Zbinden S, Fuchs S, Kornfeld H, Epstein SE, Burnett MS. CD8+ T lymphocytes regulate the arteriogenic response to ischemia by infiltrating the site of collateral vessel development and recruiting CD4+ mononuclear cells through the expression of interleukin-16. Circulation. 2006 Jan 3;113(1):118-24. doi: 10.1161/CIRCULATIONAHA.105.576702. Epub 2005 Dec 27. PMID 16380545
- [Result] Rogacev KS, Cremers B, Zawada AM, Seiler S, Binder N, Ege P, Grosse-Dunker G, Heisel I, Hornof F, Jeken J, Rebling NM, Ulrich C, Scheller B, Bohm M, Fliser D, Heine GH. CD14++CD16+ monocytes independently predict cardiovascular events: a cohort study of 951 patients referred for elective coronary angiography. J Am Coll Cardiol. 2012 Oct 16;60(16):1512-20. doi: 10.1016/j.jacc.2012.07.019. Epub 2012 Sep 19. PMID 22999728
- [Result] Gary T, Pichler M, Belaj K, Hafner F, Gerger A, Froehlich H, Eller P, Rief P, Hackl G, Pilger E, Brodmann M. Platelet-to-lymphocyte ratio: a novel marker for critical limb ischemia in peripheral arterial occlusive disease patients. PLoS One. 2013 Jul 2;8(7):e67688. doi: 10.1371/journal.pone.0067688. Print 2013. PMID 23844064
- [Result] Uzun F, Erturk M, Cakmak HA, Kalkan AK, Akturk IF, Yalcin AA, Uygur B, Bulut U, Oz K. Usefulness of the platelet-to-lymphocyte ratio in predicting long-term cardiovascular mortality in patients with peripheral arterial occlusive disease. Postepy Kardiol Interwencyjnej. 2017;13(1):32-38. doi: 10.5114/aic.2017.66184. Epub 2017 Mar 10. PMID 28344615
- [Result] Gary T, Pichler M, Belaj K, Eller P, Hafner F, Gerger A, Brodmann M. Lymphocyte-to-monocyte ratio: a novel marker for critical limb ischemia in PAOD patients. Int J Clin Pract. 2014 Dec;68(12):1483-7. doi: 10.1111/ijcp.12495. Epub 2014 Oct 31. PMID 25359092
- [Result] Teperman J, Carruthers D, Guo Y, Barnett MP, Harris AA, Sedlis SP, Pillinger M, Babaev A, Staniloae C, Attubato M, Shah B. Relationship between neutrophil-lymphocyte ratio and severity of lower extremity peripheral artery disease. Int J Cardiol. 2017 Feb 1;228:201-204. doi: 10.1016/j.ijcard.2016.11.097. Epub 2016 Nov 14. PMID 27865186
- [Result] Gary T, Pichler M, Belaj K, Hafner F, Gerger A, Froehlich H, Eller P, Pilger E, Brodmann M. Neutrophil-to-lymphocyte ratio and its association with critical limb ischemia in PAOD patients. PLoS One. 2013;8(2):e56745. doi: 10.1371/journal.pone.0056745. Epub 2013 Feb 15. PMID 23457609
- [Result] Spark JI, Sarveswaran J, Blest N, Charalabidis P, Asthana S. An elevated neutrophil-lymphocyte ratio independently predicts mortality in chronic critical limb ischemia. J Vasc Surg. 2010 Sep;52(3):632-6. doi: 10.1016/j.jvs.2010.03.067. Epub 2010 Jun 22. PMID 20573475
- [Result] Erturk M, Cakmak HA, Surgit O, Celik O, Aksu HU, Akgul O, Gurdogan M, Bulut U, Ozalp B, Akbay E, Yildirim A. Predictive value of elevated neutrophil to lymphocyte ratio for long-term cardiovascular mortality in peripheral arterial occlusive disease. J Cardiol. 2014 Nov;64(5):371-6. doi: 10.1016/j.jjcc.2014.02.019. Epub 2014 Mar 28. PMID 24685686
- [Result] Gonzalez-Fajardo JA, Brizuela-Sanz JA, Aguirre-Gervas B, Merino-Diaz B, Del Rio-Sola L, Martin-Pedrosa M, Vaquero-Puerta C. Prognostic significance of an elevated neutrophil-lymphocyte ratio in the amputation-free survival of patients with chronic critical limb ischemia. Ann Vasc Surg. 2014 May;28(4):999-1004. doi: 10.1016/j.avsg.2013.06.037. Epub 2013 Oct 27. PMID 24559786
- [Result] Zencirkiran Agus H, Kahraman S. Prognostic nutritional index predicts one-year outcome in heart failure with preserved ejection fraction. Acta Cardiol. 2020 Sep;75(5):450-455. doi: 10.1080/00015385.2019.1661139. Epub 2019 Sep 9. PMID 31498720
- [Result] Sun K, Chen S, Xu J, Li G, He Y. The prognostic significance of the prognostic nutritional index in cancer: a systematic review and meta-analysis. J Cancer Res Clin Oncol. 2014 Sep;140(9):1537-49. doi: 10.1007/s00432-014-1714-3. Epub 2014 May 31. PMID 24878931
- [Result] Lee SI, Ko KP, Choi CH, Park CH, Park KY, Son KH. Does the prognostic nutritional index have a predictive role in the outcomes of adult cardiac surgery? J Thorac Cardiovasc Surg. 2020 Jul;160(1):145-153.e3. doi: 10.1016/j.jtcvs.2019.08.069. Epub 2019 Sep 19. PMID 31627943